CLINICAL TRIAL: NCT03060031
Title: Effects of Oxytocin Administration on Social Influence Effects on Pain
Brief Title: Effects of Intranasal Oxytocin Administration on Social Influence Effects on Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Tor Wager, Director, Cognitive and Affective Neuroscience Laboratory; Professor, Department of Psychology and Neuroscience and the Institute for Cognitive Science, University of Colorado, Boulder
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: GRANT11076934
Record Dates: First submitted 2017-02-08; First posted 2017-02-23 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Pain
Keywords: Oxytocin
MeSH Terms: conditions — Pain | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oxytocin (Experimental): Each participant will undergo pain tasks after self-administration of oxytocin
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Each participant will undergo pain tasks after self-administration of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — Oxytocin intranasal administration, 40 IU, 5 puffs per nostril at 4 IU per puff delivered approximately 45 minutes prior to pain tasks.
  Other Names: Syntocinon
  Arms: Oxytocin
Drug: Placebo — Placebo intranasal administration, 5 puffs per nostril delivered approximately 45 minutes prior to pain tasks
  Arms: Placebo

SUMMARY:
This experiment will explore the joint effects of social information, social support, associative learning, and oxytocin on the development of placebo analgesia. The investigators predict that socially transmitted placebo effects will be enhanced by nasal administration of oxytocin, whereas associative learning effects on pain will not be altered by this pharmacological manipulation

DETAILED DESCRIPTION:
Background:

The placebo literature suggests that both conceptual (i.e. socially instructed beliefs) and associative learning processes are critical for the genesis of placebo effects. Several studies have performed placebo 'conditioning' (associating a sham treatment with reduced pain through repeated experience) but interfered with conceptual processing by informing subjects that the intensity of the stimulus was being lowered. This manipulation prevented the attribution of pain reductions to the placebo treatment during the learning process. These studies showed no conditioned analgesia. However, when the same 'conditioning' was performed without the verbal explanation for why the treatment seemed to work, robust placebo effects were created. Conceptual processes appear to be critical. Conversely, several studies have manipulated conceptual expectations alone, by manipulating verbal instructions, and have found markedly reduced or absent placebo analgesia on both pain report and brain event-related potentials. Learning by experience also seems to be critical.

These studies separately have led to the conclusions that 'expectancy' and 'conditioning' are each critical processes, and debates have focused on which one is the driver of placebo effects. The investigators propose another view: Both processes are critical, and they interact. Experience drives changes in value learning systems, but in any type of value learning, there is a 'credit assignment' problem, and the brain must decide which cue-outcome associations to update as a result of experience: Is the pain reduced because the treatment was effective or because the cause of pain changed? Conceptual processes fill the gap, drawing on explicit memory and generalization from similar past experiences to solve the credit assignment problem, creating analgesia if experienced relief is attributed to the treatment. This view is compatible with older information based theories of conditioning and new evidence that rats and humans alike maintain expectancies about specific outcomes and mental models of contingencies that are distinct from associative learning. In spite of dozens of published studies demonstrating effective placebo analgesia with the established paradigm the investigators use, the precise nature of the learning that occurs is unknown, because placebo analgesia has not typically been studied from a learning-systems perspective. The aim of the present study is to assess the influence of social information and associative learning on placebo analgesia.

In addition, interactions between neurochemical systems and placebo analgesia have hardly been explored, and this proposal represents a significant effort in that regard. For example, oxytocin interacts synergistically with opioids in the PAG (periaqueductal gray) (and CCK (Cholecystokinin)) to relieve pain, and in a separate literature reliably increases trust and reduces anxiety in interpersonal situations. In spite of the fact that oxytocin has been proposed as central to the placebo effect and can be administered to humans with no known subjective effects or side effects, its role in placebo analgesia has not been explored extensively. The experiment proposed here will clarify the roles of the oxytocin system and its contributions to social facilitation of analgesia, and will be instrumental in developing a systems-based model of placebo effects.

Experimental Design:

Participants will perform two tasks in each experimental session. First, they will perform a social-influence and learning task to investigate the effects of oxytocin on social instruction effects and learning on pain. Second, they will perform a social-support during pain, to test the effects of oxytocin on the pain-alleviating effects of social support during pain.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a volunteer between 18 and 40 years of age.
* If female, subject is non-lactating, not pregnant, and using a reliable contraception method
* Subject is able to read and speak English.
* Subject is able and willing to provide written informed consent.
* Subject is able to understand and follow the instructions of the investigator and understand all screening questionnaires.
* Subject is in good health.
* For participants to be eligible for all tasks of the study, the participant must have a romantic partner and be willing to bring the partner to the study session.

Exclusion Criteria:

* Tests positive on the 14 panel poly-substance urine drug screen for illicit substances (e.g., marijuana (THC), cocaine (COC), phencyclidine (PCP), amphetamine (AMP), ecstasy (MDMA), methamphetamine (Mamp), opiates (OPI), oxycodone (OXY), methadone (MTD), barbiturates (BAR), benzodiazepines (BZO), buprenorphine (BUP), tricyclic antidepressants (TCA), propoxyphene (PPX))
* Chronic Pain
* Do not have the ability to tolerate heat pain applied to the forearm
* Have temporary abnormal levels of pain
* Have score of > 19 using the Center for Disease and Epidemiology Depression Scale
* Current treatment (e.g., medications or therapy) for psychiatric disorders, including mood, anxiety, substance abuse, Attention-deficit/hyperactivity disorder (ADHD), psychosis; Neurological disorders (e.g., taking dopamine agonists for Parkinson's); Cardiovascular disease or medication (e.g., taking ACE (angiotensin-converting-enzyme) inhibitors for cardiac remodeling)
* Frequent smoking (> 5 cigarettes / day); frequent alcohol use (>14 drinks / week); frequent migraines (> 5 / month on average) or a history of neurologic disease or neuropathic pain.
* Any allergy to Oxytocin

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2019-03-05 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Change in pain expectation rating score made on a Visual Analog Scale (VAS) after administration of Oxytocin vs. Placebo | Measured during pain tasks at session 1 (within one month of screening survey completion) and 2 which will be within one week of each other.
  Self reported expectation of pain intensity using the VAS ranging from 0-100 (with 0 representing "no pain at all" and 100 representing "most intense pain imaginable (in the context of the experiment)).
Change in pain rating score made on a Visual Analog Scale (VAS) after administration of Oxytocin vs. Placebo | Measured during pain tasks at session 1(within one month of screening survey completion) and 2 which will be within one week of each other.
  Self reported pain intensity using the VAS ranging from 0-100 (with 0 representing "no pain at all" and 100 representing "most intense pain imaginable (in the context of the experiment)).
Change in pain unpleasantness rating score during hand holding and control conditions made on a Visual Analog Scale (VAS) after administration of Oxytocin vs. Placebo | Measured during pain tasks at session 1 (within one month of screening survey completion)and 2 which will be within one week of each other.
  Self reported pain unpleasantness using the VAS ranging from 0-100 (with 0 representing "no pain at all" and 100 representing "most intense pain imaginable (in the context of the experiment)).

CONTACTS AND LOCATIONS:
Overall Officials: Tor D Wager, Ph. D., Principal Investigator — University of Colorado, Boulder
Locations (1):
- Clinical Translational Research Center, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Montgomery GH, Kirsch I. Classical conditioning and the placebo effect. Pain. 1997 Aug;72(1-2):107-13. doi: 10.1016/s0304-3959(97)00016-x. PMID 9272794
- [Background] Morton DL, Watson A, El-Deredy W, Jones AK. Reproducibility of placebo analgesia: Effect of dispositional optimism. Pain. 2009 Nov;146(1-2):194-8. doi: 10.1016/j.pain.2009.07.026. Epub 2009 Aug 18. PMID 19692178
- [Background] Watson A, El-Deredy W, Iannetti GD, Lloyd D, Tracey I, Vogt BA, Nadeau V, Jones AK. Placebo conditioning and placebo analgesia modulate a common brain network during pain anticipation and perception. Pain. 2009 Sep;145(1-2):24-30. doi: 10.1016/j.pain.2009.04.003. Epub 2009 Jun 11. PMID 19523766
- [Background] Watson A, El-Deredy W, Vogt BA, Jones AK. Placebo analgesia is not due to compliance or habituation: EEG and behavioural evidence. Neuroreport. 2007 May 28;18(8):771-5. doi: 10.1097/WNR.0b013e3280c1e2a8. PMID 17471064
- [Background] Petrovic P, Kalso E, Petersson KM, Ingvar M. Placebo and opioid analgesia-- imaging a shared neuronal network. Science. 2002 Mar 1;295(5560):1737-40. doi: 10.1126/science.1067176. Epub 2002 Feb 7. PMID 11834781
- [Background] Wager TD, Rilling JK, Smith EE, Sokolik A, Casey KL, Davidson RJ, Kosslyn SM, Rose RM, Cohen JD. Placebo-induced changes in FMRI in the anticipation and experience of pain. Science. 2004 Feb 20;303(5661):1162-7. doi: 10.1126/science.1093065. PMID 14976306
- [Background] Zubieta JK, Bueller JA, Jackson LR, Scott DJ, Xu Y, Koeppe RA, Nichols TE, Stohler CS. Placebo effects mediated by endogenous opioid activity on mu-opioid receptors. J Neurosci. 2005 Aug 24;25(34):7754-62. doi: 10.1523/JNEUROSCI.0439-05.2005. PMID 16120776
- [Background] Colloca L, Tinazzi M, Recchia S, Le Pera D, Fiaschi A, Benedetti F, Valeriani M. Learning potentiates neurophysiological and behavioral placebo analgesic responses. Pain. 2008 Oct 15;139(2):306-314. doi: 10.1016/j.pain.2008.04.021. Epub 2008 Jun 6. PMID 18538928
- [Background] Kirsch I. Conditioning, expectancy, and the placebo effect: comment on Stewart-Williams and Podd (2004). Psychol Bull. 2004 Mar;130(2):341-3; discussion 344-5. doi: 10.1037/0033-2909.130.2.341. PMID 14979776
- [Background] Stewart-Williams S, Podd J. The placebo effect: dissolving the expectancy versus conditioning debate. Psychol Bull. 2004 Mar;130(2):324-40. doi: 10.1037/0033-2909.130.2.324. PMID 14979775
- [Background] Voudouris NJ, Peck CL, Coleman G. The role of conditioning and verbal expectancy in the placebo response. Pain. 1990 Oct;43(1):121-128. doi: 10.1016/0304-3959(90)90057-K. PMID 2277714
- [Background] Rescorla RA. Pavlovian conditioning. It's not what you think it is. Am Psychol. 1988 Mar;43(3):151-60. doi: 10.1037//0003-066x.43.3.151. No abstract available. PMID 3364852
- [Background] Schoenbaum G, Roesch M. Orbitofrontal cortex, associative learning, and expectancies. Neuron. 2005 Sep 1;47(5):633-6. doi: 10.1016/j.neuron.2005.07.018. PMID 16129393
- [Background] Balleine BW, O'Doherty JP. Human and rodent homologies in action control: corticostriatal determinants of goal-directed and habitual action. Neuropsychopharmacology. 2010 Jan;35(1):48-69. doi: 10.1038/npp.2009.131. PMID 19776734
- [Background] Ostlund SB, Balleine BW. Lesions of medial prefrontal cortex disrupt the acquisition but not the expression of goal-directed learning. J Neurosci. 2005 Aug 24;25(34):7763-70. doi: 10.1523/JNEUROSCI.1921-05.2005. PMID 16120777
- [Background] Balleine BW, Dickinson A. Goal-directed instrumental action: contingency and incentive learning and their cortical substrates. Neuropharmacology. 1998 Apr-May;37(4-5):407-19. doi: 10.1016/s0028-3908(98)00033-1. PMID 9704982
- [Background] Schoenbaum G, Roesch MR, Stalnaker TA, Takahashi YK. A new perspective on the role of the orbitofrontal cortex in adaptive behaviour. Nat Rev Neurosci. 2009 Dec;10(12):885-92. doi: 10.1038/nrn2753. Epub 2009 Nov 11. PMID 19904278
- [Background] Yang J, Liang JY, Li P, Pan YJ, Qiu PY, Zhang J, Hao F, Wang DX. Oxytocin in the periaqueductal gray participates in pain modulation in the rat by influencing endogenous opiate peptides. Peptides. 2011 Jun;32(6):1255-61. doi: 10.1016/j.peptides.2011.03.007. Epub 2011 Mar 23. PMID 21439337
- [Background] Ge Y, Lundeberg T, Yu LC. Blockade effect of mu and kappa opioid antagonists on the anti-nociception induced by intra-periaqueductal grey injection of oxytocin in rats. Brain Res. 2002 Feb 15;927(2):204-7. doi: 10.1016/s0006-8993(01)03346-7. PMID 11821014
- [Background] Yang J, Li P, Liang JY, Pan YJ, Yan XQ, Yan FL, Hao F, Zhang XY, Zhang J, Qiu PY, Wang DX. Oxytocin in the periaqueductal grey regulates nociception in the rat. Regul Pept. 2011 Aug 8;169(1-3):39-42. doi: 10.1016/j.regpep.2011.04.007. Epub 2011 May 3. PMID 21545817
- [Background] Reeta Kh, Mediratta PK, Rathi N, Jain H, Chugh C, Sharma KK. Role of kappa- and delta-opioid receptors in the antinociceptive effect of oxytocin in formalin-induced pain response in mice. Regul Pept. 2006 Jul 15;135(1-2):85-90. doi: 10.1016/j.regpep.2006.04.004. Epub 2006 May 19. PMID 16712978
- [Background] Kosfeld M, Heinrichs M, Zak PJ, Fischbacher U, Fehr E. Oxytocin increases trust in humans. Nature. 2005 Jun 2;435(7042):673-6. doi: 10.1038/nature03701. PMID 15931222
- [Background] Theodoridou A, Rowe AC, Penton-Voak IS, Rogers PJ. Oxytocin and social perception: oxytocin increases perceived facial trustworthiness and attractiveness. Horm Behav. 2009 Jun;56(1):128-32. doi: 10.1016/j.yhbeh.2009.03.019. Epub 2009 Apr 1. PMID 19344725
- [Background] Zak PJ, Kurzban R, Matzner WT. Oxytocin is associated with human trustworthiness. Horm Behav. 2005 Dec;48(5):522-7. doi: 10.1016/j.yhbeh.2005.07.009. Epub 2005 Aug 18. PMID 16109416
- [Background] Guastella AJ, Howard AL, Dadds MR, Mitchell P, Carson DS. A randomized controlled trial of intranasal oxytocin as an adjunct to exposure therapy for social anxiety disorder. Psychoneuroendocrinology. 2009 Jul;34(6):917-23. doi: 10.1016/j.psyneuen.2009.01.005. Epub 2009 Feb 25. PMID 19246160
- [Background] Heinrichs M, Baumgartner T, Kirschbaum C, Ehlert U. Social support and oxytocin interact to suppress cortisol and subjective responses to psychosocial stress. Biol Psychiatry. 2003 Dec 15;54(12):1389-98. doi: 10.1016/s0006-3223(03)00465-7. PMID 14675803
- [Background] Bryant RA, Hung L, Guastella AJ, Mitchell PB. Oxytocin as a moderator of hypnotizability. Psychoneuroendocrinology. 2012 Jan;37(1):162-6. doi: 10.1016/j.psyneuen.2011.05.010. Epub 2011 Jun 8. PMID 21652150
- [Background] Alvares GA, Hickie IB, Guastella AJ. Acute effects of intranasal oxytocin on subjective and behavioral responses to social rejection. Exp Clin Psychopharmacol. 2010 Aug;18(4):316-21. doi: 10.1037/a0019719. PMID 20695687
- [Background] Guastella AJ, Einfeld SL, Gray KM, Rinehart NJ, Tonge BJ, Lambert TJ, Hickie IB. Intranasal oxytocin improves emotion recognition for youth with autism spectrum disorders. Biol Psychiatry. 2010 Apr 1;67(7):692-4. doi: 10.1016/j.biopsych.2009.09.020. Epub 2009 Nov 7. PMID 19897177
- [Background] Unkelbach C, Guastella AJ, Forgas JP. Oxytocin selectively facilitates recognition of positive sex and relationship words. Psychol Sci. 2008 Nov;19(11):1092-4. doi: 10.1111/j.1467-9280.2008.02206.x. No abstract available. PMID 19076479
- [Background] Guastella AJ, Mitchell PB, Mathews F. Oxytocin enhances the encoding of positive social memories in humans. Biol Psychiatry. 2008 Aug 1;64(3):256-8. doi: 10.1016/j.biopsych.2008.02.008. Epub 2008 Mar 17. PMID 18343353
- [Background] Bartz JA, Zaki J, Ochsner KN, Bolger N, Kolevzon A, Ludwig N, Lydon JE. Effects of oxytocin on recollections of maternal care and closeness. Proc Natl Acad Sci U S A. 2010 Dec 14;107(50):21371-5. doi: 10.1073/pnas.1012669107. Epub 2010 Nov 29. PMID 21115834
- [Background] Bartz JA, Zaki J, Bolger N, Hollander E, Ludwig NN, Kolevzon A, Ochsner KN. Oxytocin selectively improves empathic accuracy. Psychol Sci. 2010 Oct;21(10):1426-8. doi: 10.1177/0956797610383439. Epub 2010 Sep 20. No abstract available. PMID 20855907
- [Background] Singer T, Snozzi R, Bird G, Petrovic P, Silani G, Heinrichs M, Dolan RJ. Effects of oxytocin and prosocial behavior on brain responses to direct and vicariously experienced pain. Emotion. 2008 Dec;8(6):781-91. doi: 10.1037/a0014195. PMID 19102589
- [Background] MacDonald E, Dadds MR, Brennan JL, Williams K, Levy F, Cauchi AJ. A review of safety, side-effects and subjective reactions to intranasal oxytocin in human research. Psychoneuroendocrinology. 2011 Sep;36(8):1114-26. doi: 10.1016/j.psyneuen.2011.02.015. Epub 2011 Mar 23. PMID 21429671